CLINICAL TRIAL: NCT03273270
Title: Effects of Neuromodulation and Rehabilitation of the Locomotor Network in Freezing of Gait
Acronym: TMS/FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS/FOG
Record Dates: First submitted 2017-08-28; First posted 2017-09-06 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease With Freezing of Gait
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): 1 Hz repetitive transcranial magnetic stimulation
  Interventions: Radiation: transcranial magnetic stimulation
- Sham TMS (Placebo Comparator): No active stimulation
  Interventions: Radiation: transcranial magnetic stimulation

INTERVENTIONS:
Radiation: transcranial magnetic stimulation — transcranial magnetic stimulation

SUMMARY:
Freezing of gait (FoG) is a common and debilitating condition in Parkinson's Disease (PD) patients. FoG is described as an episodic inability to walk, which often triggers falls, hospitalization and is an important predictor of poor quality of life. As locomotor regions degenerate in PD, gait automaticity is impaired. Patients compensate by increasing volitional control of gait, however, this adaptation has been found to worsen FoG severity. We hypothesize that increased cortical control of gait is maladaptive, and therapies to improve gait automaticity will not be effective unless cortical control of gait is reduced. The long-term goal of this project is to develop a therapeutic approach for FoG that simultaneously reduces cortical control and increases automaticity of gait. The objective is to determine the locomotor network abnormalities responsible for FoG and demonstrate how neuromodulation and rehabilitation can modulate the network. The rationale of this study is that increased connectivity between brainstem locomotor regions and cortical structures represents increased cortical governance of gait, and it can be reversed by the proposed intervention. We will accomplish this by combining a course of inhibitory rTMS (1Hz) to the cortex (supplementary motor area) with a rehabilitation protocol designed to increase gait automaticity (dual task training). We have designed a study that will carefully assess the locomotor network of freezers with resting state functional, diffusion and interleaved TMS/BOLD MRI studies, before and after intervention. Behavioral measures including gait analysis, cognitive and motor assessments will also be conducted at baseline and post treatment. The study aims to determine the effects of our intervention on the locomotor network (assessed with imaging), as well as on FoG severity as quantified through multiple markers obtained through gait analysis. At the conclusion of the study we expect to have determined the network changes central to the pathophysiology of FoG, the effects of 1Hz rTMS + rehabilitation on this network, and on FoG severity.

The relevance of this study to public health is to develop a non-invasive effective therapeutic option for one of the most debilitating and untreatable conditions affecting the lives of one million Americans suffering from PD; freezing of gait.

DETAILED DESCRIPTION:
Subjects meeting diagnostic criteria for PD and documented freezing of gait will be recruited from the MUSC Movement Disorder Clinic by clinical staff. Subjects will undergo identical imaging protocols before and after intervention. Subjects will undergo ten, 20 minute, dual task training sessions immediately following each rTMS session. Subjects will be randomized to either active rTMS + rehabilitation or rehabilitation alone at a 2:1 ratio (10 active: 5 control). The primary outcome measure will be dual task interference for turning.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting diagnostic criteria for PD and documented FoG

-

Exclusion Criteria:

* Subjects with contraindications to MRI, or TMS (no history of seizures, no metal implants in head, no pregnancy) dementia, or inability to complete the walk 30 feet in the off state without assistance will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Revuelta, DO, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TMS + Gait Training: 1 Hz repetitive transcranial magnetic stimulation
  transcranial magnetic stimulation: transcranial magnetic stimulation
- Sham TMS + Gait Training: No active stimulation
  transcranial magnetic stimulation: transcranial magnetic stimulation
Period: Overall Study
Arm/Group | Active TMS + Gait Training | Sham TMS + Gait Training
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS + Gait Training | Sham TMS + Gait Training | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (7.5) | 64.5 (8.9) | 65.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Connectivity to the Supplementary Motor Area.
Description: Change (pre vs post intervention) in resting-state fMRI connectivity (fisher z-score) of the supplemental motor area (SMA). A negative change score means there was a reduction in SMA connectivity pre to post intervention. A positive change score means there was an increase in SMA connectivity pre to post intervention.
Time Frame: pre and post intervention (within one week of completion)
Population: participant did not receive post scan due to discomfort in scanner
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Active TMS + Gait Training | Sham TMS + Gait Training
Number analyzed (Participants) | 11 | 8
z-score | -.176 (.102) | .190 (0.119)

2. Secondary Outcome: Change in New Freezing of Gait Questionnaire
Description: The new freezing of gait questionnaire is a measure of freezing severity (total score range: 0-28) wherein higher scores represent worse freezing behavior. The outcome measures represent the change in freezing of gait questionnaire score from pre to post intervention. A larger, positive value represents a greater reduction in freezing severity and a better outcome.
Time Frame: pre and post intervention (within one week of completion)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS + Gait Training | Sham TMS + Gait Training
Number analyzed (Participants) | 12 | 8
score on a scale | 4.83 (5.72) | 1.75 (3.24)

3. Secondary Outcome: Change in Dual Task Time to Turn Off
Description: The time to turn around a cone (in seconds) while dual tasking (performing a serial 7s and/or every other letter of the alphabet task) was measured while participants were in the OFF state (off of their Parkinson's medication). The assessment were performed pre to post intervention. A greater reduction in time to turn (pre versus post interverntion) is represented by a larger positive number. A larger reduction in time to turn represents a better outcome.
Time Frame: pre and post intervention (within one week of completion)
Population: Missing a pre to post measurement for one participant in the sham group
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active TMS + Gait Training | Sham TMS + Gait Training
Number analyzed (Participants) | 12 | 7
seconds | 12.05 (40.52) | 5.88 (11.94)

ADVERSE EVENTS:
Time Frame: The participants were continuously assessed for the duration of the TMS administration sessions and at pre and post intervention visits. This occurred over the time course of two weeks in which the participant was actively participating in the study.
Arm/Group | Active TMS + Gait Training | Sham TMS + Gait Training
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

LIMITATIONS AND CAVEATS:
Multiple variables were collected with gait analysis (i.e. velocity, step length, time) however, we hypothesized dual task time to turn during the OFF conditions would be most likely to change pre to post intervention. In order to minimize multiple comparisons among gait measures dual task time to turn was selected as the most important variable to detect freezing since turning and dual tasking are common triggers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03273270/Prot_SAP_000.pdf